CLINICAL TRIAL: NCT02335749
Title: CoolSculpting Treatment of the Distal Thigh
Brief Title: CoolSculpting of the Distal Thigh Study
Acronym: DST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zeltiq Aesthetics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ZA14-004
Record Dates: First submitted 2015-01-07; First posted 2015-01-12 (Estimated); Results first posted 2021-12-01 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2017-01

CONDITIONS: Body Fat Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Treatment with Small Area Applicator (Experimental): Each enrolled subject was treated on a single thigh, in the distal region.
  Interventions: Device: The ZELTIQ System

INTERVENTIONS:
Device: The ZELTIQ System — The CoolSculpting System with a Small Area Applicator will be used to deliver treatments.
  Other Names: CoolSculpting System

SUMMARY:
Evaluate the safety and efficacy of the ZELTIQ CoolSculpting System using a small area applicator for non-invasive subcutaneous fat reduction in the distal thigh.

DETAILED DESCRIPTION:
This study will investigate the use of a Small Area Applicator with the CoolSculpting device for reducing subcutaneous fat in the distal thigh. The study will evaluate the safety and effectiveness of treatments.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects > 22 years of age and < 65 years of age.
* Subject has clearly visible fat on the distal thigh, which in the investigator's opinion, may benefit from the treatment.
* Subject has not had weight change exceeding 10 pounds in the preceding month.
* Subject with body mass index (BMI) up to 30. BMI is defined as weight in pounds multiplied by 703 divided by the square of the height in inches.
* Subject agrees to maintain his/her weight (i.e., within 5% of total body weight) by not making any major changes in their diet or exercise routine during the course of the study.
* Subject has read and signed a written informed consent form.

Exclusion Criteria:

* Subject has had a surgical procedure(s) in the area of intended treatment.
* Subject has had an invasive fat reduction procedure (e.g., liposuction, mesotherapy) in the area of intended treatment.
* Subject has had a non-invasive fat reduction and/or body contouring procedure in the area of intended treatment within the past 12 months.
* Subject needs to administer, or has a known history of subcutaneous injections into the area of intended treatment (e.g., heparin, insulin) within the past month.
* Subject has a known history of cryoglobulinemia, cold urticaria, or paroxysmal cold hemoglobinuria.
* Subject has a known history of Raynaud's disease, or any known condition with a response to cold exposure that limits blood flow to the skin.
* Subject has a history of bleeding disorder or is taking any medication that in the investigator's opinion may increase the subject's risk of bruising.
* Subject is taking or has taken diet pills or supplements within the past month.
* Subject has any dermatological conditions, such as moderate to excessive skin laxity, or scars in the location of the treatment sites that may interfere with the treatment or evaluation (stretch marks is not an exclusion).
* Subject has an active implanted device such as a pacemaker, defibrillator, or drug delivery system
* Subject is pregnant or intending to become pregnant during the study period (in the next 5 months).
* Subject is lactating or has been lactating in the past 6 months.
* Subject is unable or unwilling to comply with the study requirements.
* Subject is currently enrolled in a clinical study of any other unapproved investigational drug or device.
* Any other condition or laboratory value that would, in the professional opinion of the investigator, potentially affect the subject's response or the integrity of the data or would pose an unacceptable risk to the subject.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-12-17 (Actual); Primary Completion 2015-11-09 (Actual); Study Completion 2015-11-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Bowes Dermatology Group, Miami, Florida
  - SkinCare Physicians of Chestnut Hill, Chestnut Hill, Massachusetts
  - Laser & Skin Surgery Center of New York, New York, New York
  - Nashville Centre for Laser and Facial Surgery, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment With Small Area Applicator
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All subjects who met inclusion/exclusion criteria were enrolled in the study. Once enrolled, each of the 40 subjects was treated on one distal thigh.
Arm/Group | Treatment With Small Area Applicator
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 40
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 44.6 [26.0 to 61.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 2
  African American | 1
  Hispanic | 9
  Caucasian | 28
Region of Enrollment [Number; unit: participants]
  United States | 40
Body Mass Index [Mean (Full Range); unit: kg/m^2] | 25.4 [19.7 to 30.2]

OUTCOME MEASURES:

1. Primary Outcome: Rate of Device- or Procedure-related Adverse Events
Description: The number of device- or procedure-related adverse events will be tabulated. Adverse event data are collected throughout the study period from the time of enrollment through the final follow-up visit.
Time Frame: Study enrollment through 12-week final follow-up visit, approximately 15 weeks
Population: All subjects treated with the CoolSculpting System and the Small Area Applicator were assessed for device- or procedure-lated adverse events.
Measure: Number; unit: device-or procedure-related AEs
Arm/Group | Treatment With Small Area Applicator
Number analyzed (Participants) | 40
device-or procedure-related AEs | 1

2. Primary Outcome: Proportion of Correctly Identified Photos by Blinded Reviewers
Description: Change in the treated vs. untreated areas will be assessed by observation of changes in surface contour and/or fat volume by an independent photo review of pre-treatment and post-treatment images. All reviewers will be blinded to post-treatment vs. baseline untreated area. The order in which images will be presented will be randomized; for each subject placement of the baseline, pre-treatment image will be randomized for each pair of subject images. Reviewers will be asked to select the baseline photos for each subject photo series and record selections on a data collection form.
  Note: Due to the inconsistency of site photographic practices, the photos were not reasonably evaluable and therefore the independent phot review was not conducted.
Time Frame: 12 weeks post final treatment
Population: Baseline and 12-week post-treatment photos were not reviewed by an independent panel of physicians due to inconsistencies of site photographic practices.
Units Other Than Participants: photo pairs
Arm/Group | Treatment With Small Area Applicator
Number analyzed (Participants) | 0
Number analyzed (photo pairs) | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the time of subject enrollment through the final follow-up visit, ap period of approximately 15 weeks.
Arm/Group | Treatment With Small Area Applicator
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 5/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment With Small Area Applicator (N=40)
Throat infection (Infections and infestations) | 1 (1)
Shingles (General disorders) | 1 (1) — Onset of shingles in upper arm reported.
Knee injury (General disorders) | 1 (1) — Knee injury from accidental fall was reported.
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) — Severe erythema observed on the day of treatment in the thigh area.
Bruise (Skin and subcutaneous tissue disorders) | 1 (1) — Bruise reported above treatment area of thigh. Bruise occurred after subject fell.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No